CLINICAL TRIAL: NCT01655186
Title: A Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Effects of Bardoxolone Methyl on Body Composition in Patients With Stage 4 Chronic Kidney Disease and Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IDMC recommendation for safety concerns
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-1202
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2
Keywords: Chronic Kidney Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Oral, once daily
  Interventions: Drug: Placebo
- Bardoxolone Methyl (Experimental): Oral, once daily
  Interventions: Drug: Bardoxolone Methyl

INTERVENTIONS:
Drug: Bardoxolone Methyl
  Arms: Bardoxolone Methyl
Drug: Placebo
  Arms: Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled Phase 2 safety study will assess the effect of bardoxolone methyl relative to placebo on body weight and fat mass in approximately 60 patients with stage 4 Chronic Kidney Disease (CKD) and Type 2 Diabetes Mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

1. Screening eGFR ≥ 15.0 and < 30.0 mL/min/1.73 m2; screening eGFR will be the average of the eGFR values collected during screening;
2. A history of type 2 diabetes mellitus; diagnosis must have been made at ≥ 30 years of age;
3. Male or female patients at least 30 years of age;
4. Treatment with an angiotensin converting enzyme (ACE) inhibitor and/or an angiotensin II receptor blocker (ARB) for at least 6 weeks prior to Screening Visit A and during screening. The dosage of ACE inhibitor and/or ARB must be at KDOQI goal dose (Appendix 13.4) and stable for 2 weeks prior to Screening Visit A and during screening (i.e., no change in dosage or medication);
5. Mean systolic blood pressure (SBP) must be ≤ 160 mmHg and ≥ 105 mmHg and mean diastolic blood pressure (DBP) must be < 90 mmHg during screening visits A and B;
6. Willing to practice methods of birth control (both males who have partners of childbearing potential and females of childbearing potential) during screening, while taking study drug and for at least 30 days after the last dose of study drug is ingested;
7. Serum magnesium level must be greater than or equal to 1.3 mEq/L at Screening Visit B or during a subsequent unscheduled visit during screening (serum magnesium level may be re-evaluated once during an unscheduled visit);
8. Willing and able to give written informed consent for study participation and cooperate with all aspects of the protocol including tolerating being in a closed MRI.

Exclusion Criteria:

Type 1 diabetes mellitus. If a history of diabetic ketoacidosis exists, a fasting C-peptide level must confirm type 2 diabetes; 2. Known non-diabetic renal disease (e.g., polycystic kidney disease, focal segmental glomerulosclerosis) [nephrosclerosis superimposed on diabetic kidney disease is acceptable]; Ongoing clinical investigation with evidence (e.g., unexplained hematuria or red blood cell or white blood cell casts) suggesting non-diabetic renal disease other than nephrosclerosis; 4. History of a renal transplant or a planned transplant from a living donor during the study; 5. Urine albumin/creatinine ratio (UACR) at Screening Visit B greater than 3500 mg/g; 6. Hemoglobin A1c level > 11.0% during screening; 7. Acute dialysis or acute kidney injury within 12 weeks prior to screening or during screening; 8. Clinical signs and/or symptoms of uremia and expected need for renal replacement therapy within 12 weeks following randomization, as assessed by the investigator; 9. Recently active cardiovascular disease defined as:

* Unstable angina pectoris within 12 weeks before study randomization;
* Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 12 weeks before study randomization;
* Cerebrovascular accident, including transient ischemic attack, within 12 weeks before study randomization;
* Current diagnosis of Class III or IV NYHA congestive heart failure (Appendix 13.3); 10. Clinical diagnosis of severe obstructive valvular heart disease or severe obstructive hypertrophic cardiomyopathy; 11. Atrioventricular block, 20 or 30; 12. Implanted medical device that would prevent obtaining a MRI; 13. Administration of a contrast agent that may induce nephropathy within 30 days prior to study randomization or planned during the study; 14. Systemic immunosuppression for more than 2 weeks, cumulatively, within the 12 weeks prior to randomization or anticipated need for immunosuppression during the study; 15. Total bilirubin, aspartate transaminase (AST), or alanine transaminase (ALT) level greater than the upper limit of normal (ULN) or alkaline phosphatase level greater than two times the ULN on ANY screening laboratory test result; 16. Female patients who are pregnant, intend to become pregnant during the study, or are nursing; 17. BMI < 18.5 kg/m2; 18. Weight ≥ 300 pounds; 19. Height > 6'3"; 20. Partial or total amputation of a lower extremity prior to randomization; 21. Known hypersensitivity to any component of the study drug; 22. Current history of drug or alcohol abuse, as assessed by the investigator; 23. Clinically significant infection requiring intravenous administration of antibiotics or hospitalization within 6 weeks prior to Screening Visit A or during screening; 24. Hepatitis B surface antigen positive; Diagnosis or treatment of a malignancy in the past 5 years, excluding non-melanoma skin cancer and carcinoma in situ of the cervix or a condition highly likely to transform into a malignancy during the course of the study; 26. History of bariatric surgery or planned bariatric surgery during the course of the study; 27. A clinical condition that, in the judgment of the investigator, could potentially pose a health risk to the patient while involved in the study; 28. Participation in a clinical study involving any intervention within 30 days prior to randomization, concurrent participation in such a study, or participation in a prior clinical study involving bardoxolone methyl in any form; 29. Unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09-30 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-10-31 (Actual)

PRIMARY OUTCOMES:
Mean change in body weight as measured by Dual Energy X-ray Absorptiometry (DXA) | Baseline, Weeks 12 and 24
  DXA to be done 14 days prior to or after the weeks 12 and 24 visits

SECONDARY OUTCOMES:
Mean change in fat mass as measured by Dual Energy X-ray Absorptiometry (DXA) | Baseline, Weeks 12 and 24
  DXA to be done 14 days prior to or after the weeks 12 and 24 visits
Change in visceral fat mass measured by Magnetic Resonance Imaging of the abdomen | Baseline and Week 24
  MRI to be done 14 days prior to or after the week 24 visit
Change in hepatic fat mass as measured by Magnetic Resonance Imaging of the liver | Baseline and Week 24
  MRI to be done 14 days prior to or after the week 24 visit
Change in left ventricular structure and function as measured by gated Magnetic Resonance Imaging of the heart | Baseline, Weeks 12 and 24
  MRI to be done 14 days prior to or after the weeks 12 and 24 visits
Change in gait speed | Baseline, Weeks 12 and 24
Frequency, intensity and relationship of study drug to adverse events and serious adverse events, as well as clinical, and laboratory test result abnormalities | 24 weeks

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/